CLINICAL TRIAL: NCT02246634
Title: Screening for Synchronous Metastases in Colorectal Cancer With DW-MRI.
Brief Title: Screening for Synchronous Metastases in Colorectal Cancer With DW-MRI (SERENADE)
Acronym: SERENADE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Pelican Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DOCUMAS: 17HH4153
Record Dates: First submitted 2014-09-05; First posted 2014-09-23 (Estimated); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Colorectal Neoplasms; Neoplasm Metastases; Hepatic Neoplasms
Keywords: Colorectal Neoplasms; Neoplasm Metastases; Magnetic Resonance Imaging; Diffusion Weighted MRI; Hepatic Neoplasms; Tumors; Neoplasms, Rectal
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Liver Neoplasms; Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diffusion Weighted MRI scan (Experimental): Patients who are enrolled in the study will undergo an additional diffusion weighted MRI (T2W, DWI and ADC sequences) of the liver.
  Interventions: Other: Diffusion Weighted MRI scan

INTERVENTIONS:
Other: Diffusion Weighted MRI scan — Liver metastases found on the additional DW-MRI scans will be discussed at MDT and treated according to local site policy.

SUMMARY:
Eligible patients with high risk colorectal malignancy (T3/4, spread greater than 5mm, EMVI positive) will have additional surveillance of breath hold T1, T2 and DW-MRIs (no IV contrast) post surgery six monthly for three years.

Findings of liver MRIs as reported by radiology PI will be shared with their local MDT who make decisions as appropriate, including the management of any identified liver metastases, according to local protocol.

DETAILED DESCRIPTION:
A phase II multicentre, interventional study to determine if additional staging at diagnosis with liver DW-MRI will diagnose more synchronous metastases than CT alone in patients with high risk colorectal cancer. Liver metastases found on the additional DW-MRI scans will be discussed at MDT and treated according to local policy.

ELIGIBILITY:
Inclusion Criteria:

1. Have a high risk primary colorectal malignancy
2. Have a negative CT or includes no confirmatory evidence of liver metastases
3. Is able to undergo treatment if liver metastasis is found
4. Have provided written informed consent to participate in the study
5. Be aged 16 years or over

Exclusion Criteria:

1. Have had a previous colorectal malignancy
2. Have metastatic disease
3. Have a synchronous second malignancy
4. Are contraindicated for MRI
5. Has a T3b or below low rectal tumour without EMVI or N1c

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2014-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Liver metastases found on the additional DW-MRI scans will be discussed at MDT and treated according to local site policy. | 5 years after last recruit (end of trial)
  Proportion of additional patients diagnosed with liver metastases on DW MRI compared with CT.

SECONDARY OUTCOMES:
To compare the baseline risk factors of the primary tumour against the timing and pattern of metastatic disease relapse in the liver. | 5 years after last recruit (end of trial)
  % of patients diagnosed with liver metastases according to known prognostic risk factors
To determine the sensitivity and specificity of DW-MRI as a screening method for liver lesions in patients with high risk colorectal cancer. | 5 years after last recruit (end of trial)
  % lesions suspected as metastatic on DW MRI confirmed by subsequent 'gold standard' of contrast enhanced MRI and/or surgical resection, and/or progressive enlargement of the lesion.
To describe the cancer specific disease free survival and overall survival outcomes in patients with and without liver metastases. | 6mth, 12mth, 18mth, 2yr, 3yr
  Survival and recurrence outcomes according to presence or absence of liver metastases
To characterise the patients diagnosed through screening with liver metastasis in the SERENADE study using the Fong criteria. | 5 years after last recruit (end of trial)
  Fong score of all patients with liver metastases
To describe the impact of MR screening on treatment received by patients who are diagnosed with liver metastases. | 5 years after last recruit (end of trial)
  Proportion of patients undergoing curative treatment and methods of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gina Brown, Principal Investigator — Imperial College London
Locations (13):
- United Kingdom (13):
  - Macclesfield District General Hospital, Macclesfield, Cheshire
  - Queen's Hospital, Burton-on-Trent, Derbyshire
  - Broomfield Hospital, Chelmsford, Essex
  - Royal Bolton Hospital, Bolton, Greater Manchester
  - Medway Maritime Hospital, Gillingham, Kent
  - University Hospital of South Manchester & Manchester Royal Infirmary, Wythenshawe, Manchester
  - Royal Liverpool Hospital, Liverpool, Merseyside
  - Royal Stoke University Hospital, Stoke-on-Trent, Staffordshire
  - Royal Marsden Hospital, Sutton, Surrey
  - Royal Gwent Hospital, Newport, Wales
  - George Eliot Hospital, Nuneaton, Warwickshire
  - Salisbury District Hospital, Salisbury, Wiltshire
  - Queen Alexandra Hospital, Portsmouth